CLINICAL TRIAL: NCT02915471
Title: Virtual Peer-to-peer (VP2P) Support Mentoring for Adolescents With Cancer: A Pilot Pragmatic Randomized Controlled Trial
Brief Title: Virtual Peer-to-Peer (VP2P) Support Mentoring for Adolescents With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/ NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000051755
Record Dates: First submitted 2016-09-12; First posted 2016-09-27 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Cancer
Keywords: Adolescent; Online Peer Support; Managing Cancer; Mentor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Virtual Peer-to-Peer Support Mentoring (Experimental): n addition to standard medical care, adolescents in the experimental group will receive the iP2P support program, a manualized peer-mentorship program that will provide mentoring and reinforcement by peers (young adults with cancer aged 16-25 years who have learned to function successfully with their cancer to the mentored participants).
  Interventions: Behavioral: Virtual Peer-to-Peer Support Mentoring
- Wait-list Control (No Intervention): The control group will receive usual care but without the mentorship intervention. They will be offered the iP2P support program after completion of outcome measures (T1 - to be completed online prior to randomization; T2 - at program completion).

INTERVENTIONS:
Behavioral: Virtual Peer-to-Peer Support Mentoring — The mentorship program will encourage mentored participants to develop and engage in self-management and transition skills and support their practice of these skills. The mentors will present information to mentored participants in a monitored virtual interaction using Skype for 8 weeks (10 total Skype sessions of 45 minutes each) to encourage participation in skill building tailored to their needs. All mentors will complete a paid 1.5 day training course and will be supported throughout the duration of the study (consultations with research staff to deal with unforeseen concerns). Mentored participants will complete online outcome measures prior to randomization (T1) and upon study completion (T2).
  Arms: Virtual Peer-to-Peer Support Mentoring

SUMMARY:
The overall aim of this research program is to develop and examine the impact of a Cancer virtual peer-to-peer (VP2P) Support Program on health-related quality of life (HRQL) in adolescents with cancer (AWC). In the current proposal, the feasibility of trialing the Skype-based VP2P program providing peer-support from mentors and the magnitude of program effect estimates will be evaluated in a pilot randomized control trial (RCT). This pilot RCT will enable us to refine the program and determine the appropriate sample size for a future large-scale RCT, which will compare the effectiveness of VP2P to a waitlist control group at a major Children's Oncology Group- affiliated centers in Canada and the United States.

DETAILED DESCRIPTION:
The aim of this project is to develop and examine the impact of a virtual peer support program on health outcomes and quality of life of adolescents with cancer using a waitlist randomized controlled trial. In addition to standard medical care, adolescents in the experimental group will receive a manualized peer mentorship program that will provide modelling and reinforcement by trained young adults aged 18-25 years who have learned to function successfully with their pain. Mentoring sessions consist of 10 sessions of 30-45 minute Skype calls over 8 weeks. Feasibility of the program will be measured in addition to quality of life, physical and emotional symptoms, pain coping, self-efficacy, social support, and self-management skills.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking 12-17 year olds
* Cancer diagnosis with an expected 5-year survival rate of >70% according to treating oncologist (most childhood cancer diagnoses meet this criterion1)
* Access to computer capable of using free Skype software (NB: 87% of American households had Internet access in)
* Karnofsky or Lansky performance status of 60/100 (minimal assistance needed to complete activities) as assessed by the study coordinator at the time of recruitment. The Principal Investigator and Co-Investigators (Dr. Jennifer Stinson, Dr. Nathan and Dr. Gupta) will train the study coordinator to complete Karnofsky or Lansky performance assessments.
* NB. Note that even though text messaging is part of the intervention, access to smartphones is not required. Smartphones (iPhone 6) may be loaned to participants by Dr. Stinson.

Exclusion Criteria:

* Significant cognitive impairment or major co-morbid illness as identified by their treating oncologist
* Participation in other peer support or self-management programs
* Receiving end-of-life care

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Accrual and Attrition rates | 2 months
Adherence | 2 months
  100% if calls completed over 10 weeks
Proportion of completed questionnaires | 2 months
  100% if all questions completed
Technical difficulties - developed by the investigator | 2 months
  Date, time and issue will be collected
Acceptability - semi structured interviews with AWC and mentors | 2 months
  Semi-structured interviews will be developed by the investigator

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQL) | 2 months
  Using PedsQL and its Cancer Module
Knowledge | 2 months
  Using Adolescent Cancer Knowledge Questionnaire
Perceived social support | 2 months
  Perceived Social Support from Friends
Self-efficacy | 2 months
  Generalized Self-Efficacy Sherer Scale will be used to measure self-efficacy where 1 = not true and 4 = exactly true.
  Reliability: Internal consistency is good for adolescents. α = 0.87 Validity: Evidence of good construct validity as positively correlated with Rosenberg Self-Esteem Scale.
Transition readiness | 2 months
  Transition-Q Readiness scale will be used to measure transition readiness. Reliability: Internal consistency good, α = 0.87. Test-retest reliability = 0.90 Validity: Construct validity supported by scores for transition readiness being lower for younger children (p < 0.01) and those who needed assistance completing the scale (p < 0.01). Scores were incrementally higher according to agreement with the statement, "I am ready to transfer to adult health care" (p < 0.01).
  Scale options are from 0 to 2; 0 = never, 1 = sometimes, 2 = always. A higher score refers to higher transition readiness

OTHER OUTCOMES:
Frequency and content | 2 months
  The nature (frequency and content) of the emotional, appraisal and informational support provided by mentors during VP2P sessions will be established. Data for this outcome will be collected from the audio-recorded Skype calls and text messages from each AWC-mentor dyad.
Mentor physical and emotional symptoms SF-36 physical and mental scales | 2 months
  Effect sizes for mentor physical and emotional symptoms (using SF-36 physical and mental scales)
Mentor perceived social role satisfaction - PROMIS Satisfaction with Social Roles and Activities | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada